CLINICAL TRIAL: NCT05514041
Title: A Randomized, Controlled, Double-masked, Investigator-initiated Trial to Evaluate Tear Film Quality and Stability in Subjects With Dry Eye Disease Using OC-01 (Varenicline Solution) Nasal Spray 0.03 mg as Compared to Vehicle Control Nasal Spray
Acronym: TSUNAMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stephenson Eye Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-04
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Change in Cassini surface qualifier image analysis from baseline (pre-administration) to post-administration of OC-01 (varenicline solution) nasal spray as measured by a masked evaluator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- OC-01 (varenicline solution) nasal spray 0.03 mg (Experimental): Subjects will be randomized 1:1 to be treated with the agent delivered as a 0.05 mL intranasal spray in each nostril at the following formulations
  Interventions: Drug: Varenicline solution
- Placebo nasal spray (OC-01 Vehicle Nasal Spray) (Placebo Comparator): Subjects will be randomized 1:1 to be treated with the agent delivered as a 0.05 mL intranasal spray in each nostril at the following formulations
  Interventions: Drug: Placebo nasal spray (OC-01 Vehicle Nasal Spray)

INTERVENTIONS:
Drug: Varenicline solution — OC-01 nasal spray 0.03 mg
  Arms: OC-01 (varenicline solution) nasal spray 0.03 mg
Drug: Placebo nasal spray (OC-01 Vehicle Nasal Spray) — Placebo nasal spray (OC-01 Vehicle Nasal Spray)
  Arms: Placebo nasal spray (OC-01 Vehicle Nasal Spray)

SUMMARY:
A randomized, controlled, double-masked, investigator-initiated trial to evaluate tear film quality and stability in subjects with dry eye disease using OC-01 (varenicline solution) nasal spray 0.03 mg as compared to vehicle control nasal spray.

DETAILED DESCRIPTION:
A randomized, controlled, double-masked, investigator-initiated trial to evaluate tear film quality and stability in subjects with dry eye disease using OC-01 (varenicline solution) nasal spray 0.03 mg as compared to vehicle control nasal spray.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must:

  * Provide signed written consent prior to study-related procedures
  * Be at least 22 years of age at the screening visit
  * Be literate and able to complete questionnaires independently
  * Be able and willing to use the study drug and participate in all study assessments and visits
  * Have sufficient hand strength, in the opinion of the Investigator, to be able to independently administer the study drug
  * Have provided verbal and written informed consent
  * Have an OSDI score ≥ 13,
  * Demonstrate corneal fluorescein staining (CFS) score of 2 or more in at least 1 corneal region, or a sum of 4 or more for all corneal regions, based on the National Eye Institute/Industry Workshop Scale
  * Demonstrate abnormal Cassini surface qualifier image at screening visit (at the determination of the investigator)

Exclusion Criteria:

* Subjects must not:

  1. Have undergone ocular surgery (e.g., cataract, corneal or refractive surgical procedure) within 6 months prior to the Screening/Baseline Visit
  2. Have evidence of clinically significant ocular trauma
  3. Have active ocular Herpes simplex or Herpes Zoster infection
  4. Have ocular inflammation (uveitis, iritis, scleritis, episcleritis, conjunctivitis or keratitis, with the exception of keratoconjunctivitis sicca) at the discretion of the investigator
  5. Have ocular infection (e.g., viral, bacterial, mycobacterial, protozoan or fungal infection of the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids. including hordeolum)
  6. Have severe (Grade 3 or 4) inflammation of the eyelid (e.g., blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis)
  7. Have eyelid abnormalities that significantly affect the lid function (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis)
  8. Have an ocular surface abnormality that may compromise the corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, corneal dystrophy, or the effect of any other ophthalmic medication that might in the opinion of the investigator compromise the ocular surface integrity)
  9. Have a systemic condition or disease not stabilized or judged by the Investigator to be incompatible with participation in the study or with the lengthier assessments required by the study (e.g., current systemic infection, uncontrolled autoimmune disease, uncontrolled immunodeficiency disease, history of myocardial infarction or heart disease, etc.)
  10. Have chronic or recurrent epistaxis, coagulation disorders or other conditions that, in the opinion of the Investigator, may lead to clinically significant risk of increased bleeding
  11. Have had nasal or sinus surgery (including history of application of nasal cautery) or significant trauma to these areas
  12. Have any untreated nasal infection at Visit 1
  13. Have a history of vascularized nasal polyp, severely deviated septum, chronic recurrent nosebleeds, or severe nasal obstruction
  14. Have current concomitant use of a nicotinic acetylcholine receptor agonist [Nicoderm®, Nicorette®, Nicotrol NS® (nicotine), Tabex®, Desmoxan® (cytisine), and Chantix® (varenicline)] within the previous 30 days of Visit 1 and during the treatment period.
  15. Have undergone mechanical treatment for meibomian gland dysfunction using thermal pulsation/expression (e.g., LipiFlow) or intense pulsed light (e.g., OptiLight) therapy within 6 months prior to the Screening/Baseline Visit
  16. Use topical prescription ophthalmic medications including cyclosporine and/or lifitegrast within 6 months prior to the Screening/Baseline Visit and during the treatment period
  17. Use topical ophthalmic corticosteroid therapy within 6 weeks prior to the Screening/Baseline visit and during the treatment period
  18. Use ophthalmic artificial tear drops within 2 hours prior to any of the study visits; any concurrent use of artificial tears should be continued at same frequency and with no change in brand during the treatment period
  19. Use prescription or OTC topical ophthalmic mast cell stabilizers or antihistamines within 3 days of the Screening/Baseline visit and during the treatment period (systemic agents permitted)
  20. Have a known hypersensitivity to any of the procedural agents or study drug components
  21. Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days prior to the Screening/Baseline visit and during the treatment period.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-29 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Surface qualifier image change | Day 1
  Change from baseline in Cassini surface qualifier image analysis to post-administration of OC-01 (varenicline solution) nasal spray (@15 minutes) on Day 1

SECONDARY OUTCOMES:
EDS | Day 28
  Mean change from baseline in symptom score (EDS)
Change from baseline in surface qualifier image analysis | Day 28
  Change from baseline in surface qualifier image analysis to pre-administration of varenicline solution nasal spray
Corneal fluorescein staining score | Day 28
  Mean change from baseline in corneal fluorescein staining score
TBUT | Day 28
  Mean change from baseline in fluorescein tear breakup time (TBUT)
QoL | Day 21
  Mean change from baseline in QOL questionnaire score
Tear osmolarity | Day 28
  Mean change from baseline in tear osmolarity score
VA | Day 28
  Mean change from baseline in visual acuity (logMAR)
IOP | Day 28
  Mean change from baseline in intraocular pressure

OTHER OUTCOMES:
Exploratory analysis of change in Cassini | Day 1/Day 28
  Clinical interpretation and analysis of change in Cassini surface qualifier image elapsed video
AEs | 28 days
  Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Stephenson Eye Associates, Venice, Florida, United States

IPD SHARING:
Plan to Share IPD: No